CLINICAL TRIAL: NCT05327153
Title: The Efficacy of Acceptance and Commitment Therapy (ACT) on Disease Acceptance and Quality of Life in Breast Cancer Patients: A Randomized Controlled Trial
Brief Title: The Psychology Intervention on Disease Acceptance and Quality of Life in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Song Wenjun, doctor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20220303swj0211
Record Dates: First submitted 2022-03-03; First posted 2022-04-14 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Breast cancer patients from the IPPT Breast Clinic who meet the inclusion criteria will be contacted and informed about the study and procedure. Informed consent will be obtained once the respondent agrees to participate. In the case of group psychological intervention, 8 breast cancer patients form one group, and group psychological intervention is given once a week for four weeks as part of the treatment process. The batteries of assessment were carried out at 3-time points; pre-intervention, post-intervention, and 3 months after the intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- waitlist group (Other): After the intervention of the intervention group, the waitlist group was interfered again. The batteries of assessment was same as the intervention group.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The theoretical foundation of ACT is Relational Frame Theory (RFT) based on the functional contextualism philosophy, which suggests that the main psychological problem derived verbal and cognitive interaction with environment, leading to behaviors contrary to long-term values and psychological inflexibility. The psychopathological model of ACT includes six core parts: experiential avoidance, cognitive fusion, attachment to the conceptualized self, conceptualized past and feared future, lack of value clarity, inaction.

SUMMARY:
The psychological rehabilitation of breast cancer patients plays an important role in the whole process of disease rehabilitation. In this paper, patients with breast cancer were treated with ACT group intervention for a period of four weeks to improve their disease acceptance and psychological flexibility, so as to improve their quality of life. Finally, its effect and mechanism are explored by covariance analysis and mediation analysis. The significant findings of this study will provide the quality of life changes in breast cancer patients and how did these changes happen and the moderating role of social support in the process of intervention.

DETAILED DESCRIPTION:
This is a randomized controlled trial that examines the efficacy of brief acceptance and commitment therapy by comparing the differences between ACT intervention (cases) and waitlist (control). The inclusion criteria are breast cancer patients must be 18 years old and above, early stage of breast cancer (stages 1 to 3), newly diagnosed breast cancer patients in the treatment phase and know about the illness (before and after surgery), have basic writing, reading, and verbal communication skills and volunteer to participate in this study. The exclusion criteria including patients with metastatic or recurrent breast cancer or other malignant tumors, patients had participated ACT intervention before, patients who were diagnosed with psychoses, substances abuser and people who previously exposed to chemotherapy. Respondents will be randomly recruited based on odd and even sequences. Those who are in odd sequence will be assigned into group A, and those who are in even sequence will be assigned into group B. It is stipulated that group A is the intervention group and group B is the control group. The respondents will not know in which group that they belong to ensure the single blinding process. Breast cancer patients from Breast Clinic, IPPT who met the inclusion criteria will be approached andinformed about the study and procedure will be given. Once the respondent agrees to participate, informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients must be 18 years old and above
* early stage of breast cancer (stages 1 to 3)
* newly diagnosed breast cancer patients in the treatment phase
* know about the illness (before and after surgery)
* have basic writing, reading, and verbal communication skills
* volunteer to participate in this study

Exclusion Criteria:

* breast cancer patients with more than 65 years old
* patients with metastatic or recurrent breast cancer or other malignant tumors
* patients had participated ACT intervention before
* patients who were diagnosed with psychoses, substances abuser
* people who previously exposed to chemotherapy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-10-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
To examine the efficacy of brief acceptance and commitment therapy on disease acceptance and quality of life of breast cancer patients | 10 months
  The hypothesis is that Acceptance and Commitment Therapy helps improve disease acceptance and quality of life in breast cancer patients. The study collected data through questionnaires. ANCOVA will be employed to examine the significant differences of measured variables between waitlist and intervention groups whilst controlling the covariates.

SECONDARY OUTCOMES:
The mechanism between acceptance and commitment therapy with disease acceptance and quality of life in breast cancer patients | 1 months
  The hypotheses is Acceptance and Commitment Therapy intervention can reduce the level of anxiety and depression and improve the quality of life by improving psychological flexibility and disease cognition. Meanwhile, As a way of social support, ACT intervention can moderator disease acceptance and quality of life. The study collected data through the corresponding questionnaires. Mediation analysis and moderation analysis will be computed via PROCESS macro Version 3.5 by Andrew F. Hayes.

CONTACTS AND LOCATIONS:
Overall Officials: En.Mohd Bazlan Hafidz Mukrim, phd, Principal Investigator — Setiausaha Jawatankuasa Etika Penyelidikan USM
Locations (1):
- Advanced Medical and Dental Institute Universiti Sains Malaysia, Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song W, Shari NI, Song J, Zhang R, Mansor NS, Leong Bin Abdullah MFI, Zhang Z. Effectiveness of Acceptance and Commitment Therapy (ACT) on disease acceptance for breast cancer patients: Study protocol of a randomized controlled trial. PLoS One. 2024 Nov 11;19(11):e0312669. doi: 10.1371/journal.pone.0312669. eCollection 2024. PMID 39527516